CLINICAL TRIAL: NCT01286571
Title: Bioavailability and Pharmacokinetics of 50 mg BI 135585 XX Administered as Tablet With and Without Food to Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-way Crossover Study)
Brief Title: Bioavailability and Pharmacokinetics of BI 135585 XX Administered as Tablet With and Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1283.3; 2010-022697-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — 6-(2-hydroxy-2-methylpropyl)-3-(1-(4-(1-methyl-2-oxo-1,2-dihydropyridin-4-yl)phenyl)ethyl)-6-phenyl-1,3-oxazinan-2-one

ARMS (2):
- BI 135585 (T) (Experimental): single dose per subject as tablet formulation after high fat, high caloric meal
  Interventions: Drug: BI 135585
- BI 135585 (R) (Experimental): single dose per subject as tablet formulation after an overnight fast
  Interventions: Drug: BI 135585

INTERVENTIONS:
Drug: BI 135585 — one oral single dose per subject
  Arms: BI 135585 (T)
Drug: BI 135585 — one oral single dose per subject
  Arms: BI 135585 (R)

SUMMARY:
The objective of this study is to investigate the effect of food on the relative bioavailability of a 50 mg BI 135585 XX tablet.

ELIGIBILITY:
Inclusion criteria:

- healthy male subjects

Exclusion criteria:

- Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 135585 in plasma over the time interval from 0 hours extrapolated to infinity | up to 144 hours post treatment
Maximum measured concentration of the analyte in plasma of BI 135585 in plasma over the time interval from 0 hours extrapolated to infinity | up to 144 hours post treatment

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 144 hours post treatment
Physical examination (occurrence of findings) | up to 14 days post treatment
%AUCtz-∞ (percentage of AUC0-∞ obtained by extrapolation) | up to 144 hours post treatment
tmax (time from dosing to maximum measured concentration) | up to 144 hours post treatment
λz (terminal rate constant in plasma) | up to 144 hours post treatment
t1/2 (terminal half-life of the analyte in plasma) | up to 144 hours post treatment
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 144 hours post treatment
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 144 hours post treatment
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 144 hours post treatment
Vital signs (blood pressure, pulse rate) | up to 14 days post treatment
12-lead ECG (electrocardiogram) | up to 14 days post treatment
Clinical laboratory parameters (haematology, enzymes, substrates, electrolytes, hormones of the HPA axis and the thyroid gland, and urinalysis) | up to 14 days post treatment
Incidence and severity of Adverse events | up to 14 days post treatment
Assessment of tolerability by the investigator | up to 14 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1283.3.1 Boehringer Ingelheim Investigational Site, Biberach, Germany